CLINICAL TRIAL: NCT03213301
Title: Lurbinectedin Monotherapy in Patients With Progressive Malignant Pleural Mesothelioma. A Multicenter, Single-arm Phase II Trial
Brief Title: Lurbinectedin Monotherapy in Patients With Progressive Malignant Pleural Mesothelioma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 17/16; 2017-001016-11 (EudraCT Number)
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Malignant Pleural Mesothelioma, Advanced
Keywords: Progressive Malignant Pleural Mesothelioma; Lurbinectedin; Mesothelioma; Phase II Trial
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — PM 01183

STUDY DESIGN:
Intervention Model Description: Prospective 2-stage single-arm open-label multicenter phase II trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lurbinectedin (Experimental): Lurbinectedin 3.2 mg/m2 i.v. every 3 weeks (one cycle) until progression, unacceptable toxicity or patient's withdrawal.
  Interventions: Drug: Lurbinectedin

INTERVENTIONS:
Drug: Lurbinectedin — 3.2 mg/m2 i.v. every 3 weeks
  Other Names: PM01183

SUMMARY:
Aim of this study is to provide the "proof of concept" of efficacy and tolerability of lurbinectedin monotherapy in progressive malignant mesotheliomas.

DETAILED DESCRIPTION:
Malignant mesothelioma arises from the mesothelial cells of the pleural, peritoneal or pericardial lining and is often associated with asbestos exposition. There is no cure for most malignant mesotheliomas and the scope of all three major oncological therapeutic procedures (surgery, radiotherapy and chemotherapy) is to reduce/eliminate symptoms as well as to prolong progression free survival (PFS) and/or overall survival (OS). While progressive patients are still in good health able to undertake a second-line treatment, there is no standard treatment for progressive disease.

Lurbinectedin is a novel compound structurally related to trabectedin and with similar mode of action. Pre-clinical data showed a better safety profile than trabectedin. Lurbinectedin has been already tested in different Phase I-II trials showing promising activity in ovarian, pancreatic, breast, small and non-small cell lung cancer as well as in other tumor types, with objective responses averaging 30%, disease stabilization up to 75% and having manageable toxicity. Although lurbinectedin has not been widely tested in mesotheliomas, some mesothelioma patients have been already treated with lurbinectedin where again promising activity has been observed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration and prior to any trial specific procedures
* Histologically confirmed malignant mesothelioma (all histologies are eligible)
* Progression on or after one line of platinum-based combination chemotherapy. Any previous treatment with surgery or radiotherapy is allowed
* ≤ 1 line of treatment with an immune checkpoint inhibitor
* Prior systemic treatment stopped at least 4 weeks before registration
* Measurable or evaluable disease according to the modified RECIST criteria for malignant pleural mesothelioma
* Age ≥ 18 years
* ECOG performance status ≤ 1
* Adequate bone marrow function: hemoglobin ≥ 90 g/L; absolute neutrophil count ≥ 2 x 109/L, platelet count ≥ 100 x 109/L
* Adequate hepatic function: total bilirubin ≤ 1.5 ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN); aspartate aminotransferase and alanine aminotransferase ≤ 3.0 x ULN; albumin ≥ 30 g/L
* Adequate renal function: creatinine clearance ≥ 30 mL/min/1.73, calculated according to the corrected formula of Cockcroft-Gault
* Women with child-bearing potential are using effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and during 6 months thereafter. A negative pregnancy test before registration (within 7 days) into the trial is required for all women with child-bearing potential
* Men agree not to father a child during trial treatment and during 6 months after last treatment infusion.

Exclusion Criteria:

* Known brain or leptomeningeal metastases
* History of another hematologic or primary solid tumor (except for curatively treated basal or squamous cell carcinoma of the skin, properly treated in situ malignant melanoma, in situ carcinoma of the uterine cervix or pT1-2 prostate cancer with Gleason score ≤6) within five years prior to registration
* More than one previous line of chemotherapy. Re-challenge is not allowed
* Prior treatment with lurbinectedin or trabectedin
* Treatment with any other experimental drug within 4 weeks before registration
* Concomitant use of other anti-cancer drugs, anti-cancer surgical intervention or radiotherapy except for local pain control and/or other local symptoms (e.g. pleurodesis due to dyspnea)
* Grade > 1 from any AE derived from previous treatment; alopecia any grade, grade ≤ 2 peripheral neuropathy and clinically not significant elevation of GGT grade ≤ 2 (according to the NCI-CTCAE v4.03) are allowed
* Treatment with cortisone (prednisolone > 10 mg or equivalent) for immune-mediated side effects from previous immunotherapy (if applicable)
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV), unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia)
* Severe or uncontrolled endocrinopathy due to previous immune checkpoint inhibitor treatment (if applicable)
* Known history of human immunodeficiency virus or active chronic hepatitis C or hepatitis B virus infection or any uncontrolled active systemic infection requiring intravenous antimicrobial treatment
* Known hypersensitivity to the trial drug or to any component of the trial drug
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) at 12 weeks | at 12 weeks
  PFS at 12 weeks is defined as absence of progression or death due to any cause during 12 weeks (±2 weeks) after registration.
  Patients with no tumor assessment at 12 weeks (±2 weeks) will be considered:
  * Progressed at 12 weeks, if they have no following tumor assessment within the trial (patient died, refused, started a new treatment or was lost to follow-up) or if they progress at the following tumor assessment after 12 weeks (±2 weeks).
  * Progression-free at 12 weeks, if they do not progress at the following tumor assessment after 12 weeks (±2 weeks).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of registration until the date of first documented relapse or progression according to the modified RECIST criteria for malignant pleural mesothelioma or date of death from any cause, whichever came first, assessed up to 30 months.
  PFS is defined as time from registration to one of the following events, whichever occurs first:
  * Relapse or progression according to the modified RECIST criteria for malignant pleural mesothelioma
  * Death due to any cause Patients not experiencing an event will be censored at the date of last evaluable tumor assessment before starting a subsequent treatment, if any.
Objective response (OR) | From date of registration until the date of treatment discontinuation for any cause, assessed up to 30 months.
  OR is defined as complete response (CR) or partial response (PR) achieved by the patient during trial treatment. Tumor response will be evaluated according to the modified RECIST criteria for malignant pleural mesothelioma.
  Patients without any tumor assessment during trial treatment will be regarded as having a non-evaluable response (NE) and shall be considered as failures for this endpoint.
Disease control (DC) at 12 weeks | at 12 weeks: From date of registration until 14 weeks after.
  DC is defined as CR, PR or stable disease (SD) for at least 12 weeks achieved by the patient during trial treatment. Tumor response will be evaluated according to the modified RECIST criteria for malignant pleural mesothelioma.
Overall survival (OS) | From date of registration until the date of death from any cause, assessed up to 30 months.
  OS is defined as time from registration until death due to any cause. Patients alive or lost to follow-up will be censored at the last date they were known to be alive.
Time to treatment failure (TTF) | From date of registration until the date of treatment discontinuation for any cause, assessed up to 30 months.
  TTF is defined as time from registration until treatment discontinuation due to any reason (unacceptable toxicity, patient refusal, progression, death or any other event that determines the termination of the trial treatment).
  Patients not experiencing an event will be censored at the date of their last available assessment or visit.

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Metaxas, MD, Study Director — Kantonsspital Graubünden, Chur; Roger von Moos, Prof, Study Chair — Kantonsspital Graubünden, Chur; Miklos Pless, MD, Study Chair — Kantonsspital Winterthur KSW; Federica Grosso, MD, Study Chair — SS. Antonio e C. Arrigo Hospital Alessandria (Italy)
Locations (8):
- Italy (2):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Istituto Clinico Humanitas, Rozzano
- Switzerland (6):
  - Kantonsspital Baden, Baden
  - IOSI Ospedale Regionale di Bellinzona e Valli, Bellinzona
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital St.Gallen, Sankt Gallen
  - Regionalspital Thun, Thun
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metaxas Y, Fruh M, Eboulet EI, Grosso F, Pless M, Zucali PA, Ceresoli GL, Mark M, Schneider M, Maconi A, Perrino M, Biaggi-Rudolf C, Froesch P, Schmid S, Waibel C, Appenzeller C, Rauch D, von Moos R; Swiss Group for Clinical Cancer Research (SAKK). Lurbinectedin as second- or third-line palliative therapy in malignant pleural mesothelioma: an international, multi-centre, single-arm, phase II trial (SAKK 17/16). Ann Oncol. 2020 Apr;31(4):495-500. doi: 10.1016/j.annonc.2019.12.009. Epub 2020 Jan 16. PMID 32085891